CLINICAL TRIAL: NCT01102179
Title: Prevalence of Vitamin D Insufficiency and Deficiency in Chronic Kidney Disease Patients in Singapore
Brief Title: Vitamin D Insufficiency and Deficiency in Chronic Kidney Disease (CKD) Patients in Singapore
Status: Completed | Type: Observational
Sponsor: National University of Singapore (Other)
Collaborators: National Kidney Foundation, Singapore (Other)
Responsible Party: Dr. Priscilla How, National University Singapore/National University Hospital
Other Study IDs: DSRB Domain E/09/643
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-10

CONDITIONS: Stage 2-5 Chronic Kidney Disease; Predialysis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic kidney disease: All patients with stage 2-5 (pre-dialysis) chronic kidney disease
  One-time blood draw (10 ml)

SUMMARY:
Vitamin D insufficiency and deficiency is common in chronic kidney disease (CKD) patients and is associated with elevated parathyroid hormone (PTH) concentration and mineral and bone disorder (MBD). There is also increasing evidence to show that these abnormalities increase cardiovascular morbidity and mortality in CKD patients. There is a need for early identification of vitamin D insufficiency/deficiency in CKD patients to prevent its long-term complications. However, the vitamin D status of CKD patients in Singapore has not been well described. The purpose of this study is to assess the vitamin D status of predialysis CKD patients in a tertiary academic teaching hospital in Singapore, and its association with parameters for MBD. Predialysis patients from the outpatient renal clinic at the National University Hospital (NUH) will be recruited into this study. Blood samples from the patients will be collected after an overnight fast to determine their serum 25(OH)D, creatinine, phosphorus, calcium, albumin and i-PTH concentrations. These parameters will be compared among patients in various stages of CKD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 21 years of age or older
* CKD stage 2 to 5 (who are not on dialysis): CKD stage 2: eGFR 60-89ml/min/1.73m2, stage 3: eGFR 30-59ml/min/1.73m2, stage 4: eGFR 15-29 ml/min/1.73m2, stage 5 eGFR <15 ml/min/1.73m2)
* Not receiving over-the-counter or prescription vitamin D therapy
* On a stable dose of phosphate binder (if any) for at least 1 month prior to the study

Exclusion Criteria:

* History of liver and chronic inflammatory diseases, primary hyperparathyroidism and malignancies
* Use of corticosteroids, anticonvulsants or vitamin D compounds
* Use of an investigational agent within 30 days of study entry

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage 2-5 chronic kidney disease who are not on dialysis
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2010-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Vitamin D 25(OH)D levels | baseline
  Vitamin D levels are only measured at one time point i.e. at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla P How, Pharm.D., Principal Investigator — National University of Singapore/National University Hospital
Locations (1):
- National University Hospital, Singapore, Singapore